CLINICAL TRIAL: NCT02418988
Title: Multicenter, Open-labeled, Controlled Phase II Study: Trans-catheter Chemo-embolization Combined With rAd-p53 Gene Injection in Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Trans-catheter Chemo-embolization Combined With rAd-p53 Gene Injection in Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: rAd-p53-H14006
Record Dates: First submitted 2015-03-25; First posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: Advanced Adult Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TACE plus rAd-p53 (Experimental): TACE plus rAd-p53 artery injection'
  Interventions: Drug: TACE plus rAd-p53 artery injection
- TACE (Active Comparator): TACE will be applied alone
  Interventions: Drug: TACE

INTERVENTIONS:
Drug: TACE plus rAd-p53 artery injection — Trans-catheter chemo-embolization (TACE) with rAd-p53 injection will be given every 21 days
  Other Names: no other name
  Arms: TACE plus rAd-p53
Drug: TACE — Trans-catheter chemo-embolization (TACE) without rAd-p53 injection will be given every 21 days
  Other Names: no other name
  Arms: TACE

SUMMARY:
Treatment options for advanced hepatocellular carcinoma (HCC) are limited due to patients' poor condition, advanced tumor, concomitant intra- and extra-liver diseases, and resistance to both chemo- and radio-therapy. Trans-catheter embolization (TAE) or Trans-catheter chemo-embolization (TACE) is the most widely used locoregional treatment for advanced HCC. But no solid evidences support the beneficial effect of the chemotherapy in TACE. Many advanced HCC patients also can't tolerate the locoregional chemotherapy. The p53 gene has multiple anticancer functions and does not have any of the immune-inhibitory effects of chemo- or radio-therapy. The objectives of this study are to investigate the efficacy and safety usingTAE plus recombinant adenoviral human p53 gene (rAd-p53) in treatment of advanced HCC.

DETAILED DESCRIPTION:
Study design: multicenter, open-labeled, active-controlled phase II study

Study treatments: TACE combined with rAd-p53 injection vs.TACE. The treatments are given once per 21 days until the disease progression. For the experiment group, 2 X 1000,000,000,000 viral particles of rAd-p53 will be injected into the embolization artery.

Study objectives: efficacy and safety of the study treatments

Study endpoints: safety (adverse events, vital signs, lab tests, ECG and physical examination) and efficacy (progression-free survival, overall survival, and ECOG PS)

ELIGIBILITY:
Inclusion Criteria:

1. histopathologically diagnosed HCC;
2. unresectable;
3. over 18 years old;
4. with an Eastern Cooperative Oncology Group (ECOG) score of 0-2;
5. with Barcelona Clinic Liver Cancer (BCLC) Stage of B or C;
6. with Child-Pugh score A or B;
7. with normal tests of hemogram, blood coagulation, liver and kidney function; 8. signed the informed consent form.

Exclusion Criteria:

1. Serious blood coagulation disorder, bleeding tendency, platelet < 6 * 1000000000/L;
2. have serious heart, lung function abnormalities or severe diabetes patients;
3. active infection;
4. liver function Child-Pugh grade C;
5. secondary and diffuse hepatocellular carcinoma patients;
6. extensive metastasis;
7. severe atherosclerosis;
8. AIDS patients;
9. serious thrombotic or embolic events within 6 months;
10. renal insufficiency requiring hemodialysis or peritoneal dialysis;

12. pregnant or lactating women;

13. mental disorder or disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | tumor assessment will be performed every 6 weeks from starting study treatment to death or 2 years later
  overall survival

SECONDARY OUTCOMES:
safety as assessed by adverse events, vital sign, lab tests, ECG and physical examination | from the first study treatment to the 30 days after the last treatment (on an average of 6 months from the start treatment)
  safety variables: adverse events, vital sign, lab tests, ECG and physical examination
progression-free survival | tumor assessment will be performed every 6 weeks from starting study treatment to disease progression or 2 years later
  time to disease progression (death or progression), or censored

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of the Fourth Military Medical University, Xi’an, Shanxi, China